CLINICAL TRIAL: NCT06215287
Title: Survey to Assess Physicians' Knowledge of Exjade Posology and Biological Monitoring Recommendations as Described in the Educational Materials
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CICL670A2429; EUPAS104950 (Other: EU PAS registry)
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Chronic Iron Overload
Keywords: Physician Survey,; PAS,; Deferasirox

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Exjade Prescribers/HCP receiving Educational Materials: HCPs prescribing Exjade in the EU/EEA provided with Exjade Educational Materials
  Interventions: Other: Physician survey

INTERVENTIONS:
Other: Physician survey — Survey to assess physicians' knowledge of Exjade posology and biological monitoring recommendations as described in the Educational Materials

SUMMARY:
The objective of this survey is to assess the knowledge of HCPs in relation to the recommended posology and biological monitoring for Exjade, based on the current locally valid Exjade educational materials (including the physician's reference checklist)

ELIGIBILITY:
Inclusion Criteria:

Physicians will be required to meet all of the following inclusion criteria:

* Must provide consent for participation
* Must spend ≥50% of time in direct patient care
* Have treated patients with transfusional iron overload or non-transfusion-dependent thalassemia with chelation therapy during the last 12 months.
* Have prescribed Exjade and/or generic deferasirox within the last 12 months.

Exclusion Criteria:

Physicians meeting the following criterion will not be eligible to take the survey:

• Currently employed by a pharmaceutical company, health care company, market research company, advertising agency, or government agency involved in pharmaceutical research or marketing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exjade (deferasirox) prescribers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Mean percentage of correct responses related to knowledge of posology and biological monitoring recommendations as described in the Exjade EU Summary of Product Characteristics (SmPC) | Through study completion, an average of 6 months.
  The primary endpoint is a composite endpoint based on the percentages of HCPs with correct responses to all questions included in the composite regarding the below information:
  * Administration and dosing of Exjade (deferasirox) FCT
  * Biological monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No